CLINICAL TRIAL: NCT02094066
Title: The Effects of High Doze Tranexamic Acid Application on Hemorrhage, Blood Transfusion, Fibrin Degradation Products, and Kidney Functions for Total Hip Arthroplasty
Brief Title: The Effect of Tranexamic Acid for Total Hip Arthroplasty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, seher orbay yasli, resident, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012/683
Record Dates: First submitted 2014-03-19; First posted 2014-03-21 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Hemorrhage
Keywords: tranexamic acid; total hip arthroplasty
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- tranexamic acid (Active Comparator): preoperative ıv 50 mg/kg tranexamic acid infusion at 45 minutes
  Interventions: Drug: tranexamic acid
- serum physiologic (Sham Comparator): preoperative 100 cc serum physiologic
  Interventions: Drug: serum physiologic

INTERVENTIONS:
Drug: tranexamic acid — preoperative ıv 50 mg/kg tranexamic acid infusion at 45 minutes
  Other Names: lysteda
  Arms: tranexamic acid
Drug: serum physiologic — preoperative 100 cc ıv serum physiologic
  Arms: serum physiologic

SUMMARY:
The aim of this study is to investigate the effects of tranexamic acid on hemorrhage, blood transfusion, fibrin degradation products and kidney functions for total hip arthroplasty.

DETAILED DESCRIPTION:
Orthopedic surgery may be associated with substantial blood loss requiring transfusion of erythrocytes.Transfusion of allogeneic erythrocytes is not free of adverse events and has been associated with transmission of infectious diseases, increased postoperative bacterial infection, immune sensitization, and transfusion related acute lung injury. Measures taken to allay concerns about the safety of blood transfusions have translated into the increasing cost of allogeneic blood units. Blood banks regularly undergo blood shortages. For these reasons, there is a need to reduce allogeneic blood transfusions. A number of effective interventions have been developed, such as preoperative autologous donation, cell salvage, or the use of erythropoietin. Pharmacologic agents such as aprotinin, tranexamic acid, or epsilon-aminocaproic acid (EACA) could reduce perioperative blood loss by interfering with fibrinolysis.

ELIGIBILITY:
Inclusion Criteria:

* ASA 2-3
* 18-75 age
* total hip arthroplasty surgery
* regional anesthesia

Exclusion Criteria:

* allergies to drug
* liver and kidney failure
* ischemic heart disease
* coagulopathy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-06 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
hemorrhage | intraoperative
  the amount of bleeding in aspirator and sponges

SECONDARY OUTCOMES:
erythrocyte transfusion | intraoperative and postoperative 3 days

CONTACTS AND LOCATIONS:
Overall Officials: seher orbay yasli, resident, Principal Investigator — Erciyes university medicine faculty
Locations (1):
- Erciyes univercity medicine faculty, Kayseri, Turkey (Türkiye)